CLINICAL TRIAL: NCT01481961
Title: Feasibility Study: Cognitive Effect of Repetitive Transcranial Magnetic Stimulation (rTMS)on add-on in Patients With Early Alzheimer's Disease
Brief Title: Study of Repetitive Transcranial Magnetic Stimulation (rTMS) as add-on Treatment for Early Alzheimer's Disease
Acronym: ALSTIMAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Vandel, MD PhD (Other)
Collaborators: Neurology department of CHU Besancon (Dr Rumbach L, Dr Berger E, Dr Galmiche J) (Unknown); Memory Center of Research and Resources (MCRR) of Besancon (Dr Magnin E) (Unknown); Rapid-fr network (Dr Galmiche J) (Unknown); Clinical Investigation Centre for Innovative Technology Network (Network); Funding by French Internal Project Call for Clinical Research(2010-A00659-30) (Unknown)
Responsible Party: Sponsor-Investigator, Pierre Vandel, MD PhD, PU PH, Centre Hospitalier Universitaire de Besancon
Organization: Centre Hospitalier Universitaire de Besancon (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALSTIMAG
Record Dates: First submitted 2011-11-23; First posted 2011-11-30 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Alzheimer's Disease; Cognition Disorders
Keywords: Alzheimer's disease; rTMS; cognition
MeSH Terms: conditions — Alzheimer Disease; Cognition Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rTMS arm (Experimental)
  Interventions: Procedure: repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Procedure: repetitive Transcranial Magnetic Stimulation (rTMS) — After locating the left DLPFC, treatment with active rTMS will be directed by 20-minute session during which pulse trains of 5 seconds of 10 Hz spaced 25 seconds (2 trains of pulses per minute or 40 pulse trains per session). Treatment will occur 2 sessions per day during 5 days per week. Subjects will be monitored during rTMS for any side effects or adverse events.

SUMMARY:
The aim is to examine the effect of Repetitive Transcranial Magnetic Stimulation (rTMS) applied at the anodic left Cortex DorsoLateral PreFrontal (CDLPF) of patients with early Alzheimer's disease (AD).

This study included 15 patients treated with rTMS and whose medication reference is stabilized for 3 months by IAChE. Patients with early AD or related disease will be selected in the MCRR of Besançon and the psychiatric department of the University Hospital of Besançon. After giving informed consent, patients will be evaluated by a psychiatrist using the Mattis Clinical Demantia Rate (CDR), the Hamilton Depression Rating Scale (HDRS), State-Trait Anxiety Inventory (STAI), Beck Depression Inventory (BDI) and Hamilton Anxiety Scale (HAMA). The complete assessment takes 40 minutes. A second evaluation will be realized by a neuropsychologist takes around 120 minutes using Mattis CDR, Grober Free and Cued Selective Reminding Test, Trail Making Test (TMT), Crossing of Test (COT), Isaacs Set Test (STI) , Clock-Drawing Test (COT), Signoret's Battery of Cognitive Efficacy (BEC96), Rey-complex figure test-copy and Picture naming 80 items test (DO80).

Each rTMS session runs 20 minutes during which pulse trains of 5 seconds of 10 Hz spaced 25 seconds (2 trains of pulses per minute or 40 pulse trains per session) will be delivered. A psychometric assessment will be conducted again at the end of treatment week and one month after stopping treatment. A neuropsychometric assessment will be conducted one month after stopping the treatment. Scales of comfort and acceptability will also be proposed to the patient to determine whether any gene is caused by this treatment. Moreover a questionnaire will be proposed to the caregivers (at baseline, at the end of the treatment and 1, 2, 3 and 4 weeks after stopping the sessions) using Resource Utilisation Dementia (RUD), Apathy Inventory (AI), Activities of Daily Living (ADL) scale, Instrumental Activities of Daily Living (IADL) scale, Quality of Life in Alzheimer's disease (QoL-AD) scale, Questionnaire of recent change of the personality (CP6).

The population of this study will be comprised of patients between 60 to 85 years-old with early Alzheimer's characterized according to NINCDS-ADRADA criteria. These patients will be recruited on a voluntary basis, after notification and consent in the research center. This study was conducted over a period of 15 months.

ELIGIBILITY:
Inclusion Criteria:

* subject diagnosed with early Alzheimer's disease or related diseases according to NINCDS-ACDRADA criteria.
* subject under treatment by IAChE for at least 3 months.
* CDR score ≤ 2
* psychotropic treatments are tolerated if they were administered and unchanged for at least 3 months

Exclusion Criteria:

* CDR > 2
* subjects diagnosed with psychiatric disorder (depression according to DSM-IV criteria, bipolar disorder, schizophrenia, addiction)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
changes in MMSE (Mini Mental State Examination) | baseline, 1wk, 4wk
  The changes in MMSE will constitute the major research outcome measure used to assess response to rTMS.

SECONDARY OUTCOMES:
changes in HDRS (Hamilton Depression Rating Scale) | baseline, 1wk, 4wk
changes in STAI (State-Trait Anxiety Inventory) | baseline, 1wk, 4wk
changes in BDI (Beck Depression Inventory) | baseline, 1wk, 4 wk
changes in HAMA (Hamilton Anxiety Scale) | baseline, 1 wk, 4 wk
changes in Mattis DRS (Dementia Rating Scale) | baseline, 1 wk, 4 wk
changes in CDR (Clinical Dementia Rate) | baseline, 1 wk, 4 wk
changes in Grober Free and Cued Selective Reminding Test | baseline, 4 wk
changes in TMT (Trail Making Test) | baseline, 4 wk
changes in COT (Crossing Of Test) | baseline, 4 wk
changes in IST (Isaacs Set Test) | baseline, 4 wk
changes in CDT (Clock-Drawing Test) | baseline, 4 wk
changes in Signoret's Battery of Cognitive Efficacy (BEC96) | baseline, 4 wk
changes in Rey-complex figure test-copy | baseline, 4 wk
changes in Picture naming 80 items test (DO80) | baseline, 4 wk
changes in RUD (Resource Utilisation Dementia) | baseline, at the end of treatment, 1wk, 2 wk, 3 wk, 4 wk
changes in AI (Apathy Inventory) | baseline, at the end of treatment, 1wk, 2 wk, 3 wk, 4 wk
changes in ADL (Activities of Daily Living) | baseline, at the end of treatment, 1wk, 2 wk, 3 wk, 4 wk
changes in IADL (Instrumental Activities of Daily Living) | baseline, at the end of treatment, 1wk, 2 wk, 3 wk, 4 wk
changes in QoL-AD (Quality of Life in Alzheimer's Disease) | baseline, at the end of treatment, 1wk, 2 wk, 3 wk, 4 wk
changes in CP6 (Questionnaire of recent change in personnality) | baseline, at the end of treatment, 1wk, 2 wk, 3 wk, 4 wk

CONTACTS AND LOCATIONS:
Overall Officials: Pierre VANDEL, Prof, Principal Investigator — Psychiatry clinical department - CHU Besançon
Locations (1):
- Psychiatric Department of CHU of Besancon, Besançon, France

REFERENCES:
- [Result] Haffen E, Chopard G, Pretalli JB, Magnin E, Nicolier M, Monnin J, Galmiche J, Rumbach L, Pazart L, Sechter D, Vandel P. A case report of daily left prefrontal repetitive transcranial magnetic stimulation (rTMS) as an adjunctive treatment for Alzheimer disease. Brain Stimul. 2012 Jul;5(3):264-266. doi: 10.1016/j.brs.2011.03.003. Epub 2011 Mar 30. No abstract available. PMID 22037125